CLINICAL TRIAL: NCT00001355
Title: Detection and Characterization of Host Defense Defects
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: University of Miami (Other); University of South Florida (Other)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 930119; 93-I-0119
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-30

CONDITIONS: Immune Defects
Keywords: Immune Deficiency; Infection; Phagocytes; Cytokines; Genetics; Natural History
MeSH Terms: conditions — Immunologic Deficiency Syndromes; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Volunteer: Healthy Volunteer to serve as controls
- Patient: Patients known to have or suspected of having an immune defect significantly or primarily involving the phagocytes
- Patient Relatives: blood relatives of patients

SUMMARY:
This protocol is designed to evaluate selected patients with documented recurrent or unusual infections and their family members for clinical and laboratory correlates of immune abnormalities. It allows long term follow up of patients with host defense defects and permits the periodic study of their blood, urine, saliva, skin, stool and vaginal specimens or wound drainage from such patients or their family members for medically indicated purposes and research studies related to understanding the genetic and biochemical bases of these diseases. This protocol may help provide patients and materials for the development of therapies for these diseases.

This study will:

1. Determine the biochemical and genetic causes of inherited immune diseases affecting phagocytes (white blood cells that defend against bacterial and fungal infections)
2. Try to develop better ways to diagnose and treat patients with these diseases, and to prevent, diagnose and treat their infections

Patients and family members may undergo the following procedures:

* A personal and family medical history, physical examination and other procedures, which may include various blood tests; urinalysis; saliva collection; imaging studies such as chest X-ray, computed tomography (CT) or magnetic resonance imaging (MRI); and lung function studies, dental examination or eye examinations, if medically indicated.
* Patients who have draining wounds will have fluid collected from these wounds for biochemical study.
* Tissues removed as part of medical care, such as pieces of lung, liver, or teeth, or biopsies of these tissues will be studied.
* Patients who have an immune problem that investigators wish to study further will be asked to return to NIH for follow-up visits at irregular intervals, but at least every 6 months. The visits will include an updated medical history, examination directed at the particular medical problem related to the immune disorder, follow-up of abnormal tests or treatment, and collection of blood, saliva, urine, or wound fluid for study.
* Patients may have genetic testing and must be willing to have specimens stored for future research.
* Family members will have a medical history, saliva or urine collection, and chest X-ray or other imaging study, if medically indicated.
* Normal volunteers who have had tissue biopsies or pieces of tissue removed as part of medical care, such as pieces of lung, liver, or teeth, will have these tissues studied.
* NIH does not cover the cost of the initial screening visit for travel or lodging. A financial assessment may determine if the patient is eligible for financial assistance. This study does not enroll children under the age of 2.
* Patients will be asked to obtain their medical records, previous test results, or imaging studies prior to the first visit.

DETAILED DESCRIPTION:
This protocol is designed to evaluate selected patients with documented recurrent or unusual infections and their family members for clinical and in vitro correlates of immune abnormalities. It will also allow long term follow up of patients with host defense defects and permit us to periodically obtain blood, urine, saliva, skin, other excess biopsy tissue, breast milk, stool and vaginal specimens or wound drainage from such patients or their family members for medically indicated purposes and research studies related to understanding the genetic and biochemical bases of these diseases. This protocol may help provide patients and materials for the development of therapies for these diseases in the future.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients known to have or suspected of having an immune defect significantly or primarily involving the phagocytes will be eligible for enrollment, as well as their blood relatives. Such syndromes include but are not limited to those listed above. Eligibility will not be limited based on sex, race, or disability. Patients or patient relatives must be over 1 month of age.

The patient and patient relative cohorts will include the following special populations:

* Children: Children are included in this study because immune defects may present in early childhood, and early diagnosis or characterization may benefit subjects.
* Decisionally impaired adults: Patients and patient relatives will be able to provide informed consent for themselves or if they lack the capacity to provide informed consent, the study team will obtain consent from the legally authorized representative. Patients with underlying immune disorders, autoimmune phenomena or severe infections may sometimes present with delirium, encephalopathy, or coma and are therefore unable to provide informed consent. Excluding patients who are unable to provide consent could adversely impact patient access to medical therapy at the NIH as well as adversely impact research recruitment. Excluding patients unable to provide consent would also essentially prohibit us from evaluating patients at higher risk for adverse outcomes and therefore skew our understanding of disease. Similarly, enrolled patient subjects who lose the ability to provide ongoing consent during study participation may continue in the study. The risks and benefits of participation for subjects unable to consent should be identical to those described for less vulnerable patients. The process for obtaining consent for these individuals is described below.

Healthy volunteers will be healthy adults between the age of 18 and 80 years of either sex, and they must be able to provide informed consents for themselves.

EXCLUSION CRITERIA:

The presence of an acquired abnormality which leads to immune defects, such as HIV, cytotoxic chemotherapy or malignancy, could be grounds for possible exclusion if, in the opinion of the investigator, the presence of such disease process interfered with evaluation.

Individuals with dementia that impairs obtaining informed consent are excluded from enrolling as healthy volunteers, although such subjects may enroll in the patient or relative cohorts if consent can be obtained as described below.

Ages: 1 Month to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants known to have or suspected of having an immune defect and their blood relatives are eligible for enrollment.@@@
Sampling Method: Non-Probability Sample
Enrollment: 3600 (Estimated)
Dates: Start 1993-09-01 (Actual)

PRIMARY OUTCOMES:
Improved disease if either normalization or sustained improvement is observed. | Complete withdrawal from steroid or sustained reduction to low dose antimicrobials or immune modulators.
  The primary endpoint of this study will be determination of a discrete diagnosis of an infecting agent, an underlying susceptibility trait, or both.

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Holland, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share human data generated in this study for future research as follows:@@@@@@@@@@@@ (Summation)Identified data in the Biomedical Translational Research Information System (BTRIS, automatic for activities in the NIH CC).@@@@@@@@@@@@ (Summation)De-identified or identified data with approved outside collaborators under appropriate agreements.@@@@@@@@@@@@ (Summation)Data sharing may be complicated or limited in certain cases by contractual obligations or agreements with outside collaborators, such as cooperative research and development agreements, clinical trial agreements, other restraints, etc.
Supporting Information: SAP
Time Frame: IPD and supporting information will be available after completion of the study. No end date.
Access Criteria: Data will be shared through:@@@@@@@@@@@@ (Summation)BTRIS (automatic for activities in the NIH CC).@@@@@@@@@@@@ (Summation)Approved outside collaborators under appropriate individual agreements.@@@@@@@@@@@@ (Summation)Publication and/or public presentations.@@@@@@@@@@@@Data might be shared before publication.@@@@@@@@@@@@The PI will review all requests for sharing data.

REFERENCES:
- [Derived] Donko A, Sharapova SO, Kabat J, Ganesan S, Hauck FH, Bergerson JRE, Marois L, Abbott J, Moshous D, Williams KW, Campbell N, Martin PL, Lagresle-Peyrou C, Trojan T, Kuzmenko NB, Deordieva EA, Raykina EV, Abers MS, Abolhassani H, Barlogis V, Milla C, Hall G, Mousallem T, Church J, Kapoor N, Cros G, Chapdelaine H, Franco-Jarava C, Lopez-Lerma I, Miano M, Leiding JW, Klein C, Stasia MJ, Fischer A, Hsiao KC, Martelius T, Seppanen MRJ, Barmettler S, Walter J, Masmas TN, Mukhina AA, Falcone EL, Kracker S, Shcherbina A, Holland SM, Leto TL, Hsu AP. Clinical and functional spectrum of RAC2-related immunodeficiency. Blood. 2024 Apr 11;143(15):1476-1487. doi: 10.1182/blood.2023022098. PMID 38194689
- [Derived] Schindler MK, Pittaluga S, Enose-Akahata Y, Su HC, Rao VK, Rump A, Jacobson S, Cortese I, Reich DS, Uzel G. Haploinsufficiency of immune checkpoint receptor CTLA4 induces a distinct neuroinflammatory disorder. J Clin Invest. 2020 Oct 1;130(10):5551-5561. doi: 10.1172/JCI135947. PMID 32955488
- [Derived] Burbelo PD, Browne SK, Sampaio EP, Giaccone G, Zaman R, Kristosturyan E, Rajan A, Ding L, Ching KH, Berman A, Oliveira JB, Hsu AP, Klimavicz CM, Iadarola MJ, Holland SM. Anti-cytokine autoantibodies are associated with opportunistic infection in patients with thymic neoplasia. Blood. 2010 Dec 2;116(23):4848-58. doi: 10.1182/blood-2010-05-286161. Epub 2010 Aug 17. PMID 20716769
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1993-I-0119.html